CLINICAL TRIAL: NCT02261896
Title: Multicenter, Randomized and Double-blinded Clinical Trial on the Use of Antibiotic Prophylaxis for EUS Guided FNA of Pancreatic Cystic Lesions
Brief Title: Antibiotic Prophylaxis for Endoscopic Ultrasound Guided Fine Needle Aspiration of Pancreatic Cystic Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IIBSP-CIP-2013-166
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Cystic Lesion
Keywords: cyst; pancreatic cyst; EUS-FNA; antibiotic prophylaxis
MeSH Terms: conditions — Cysts; Pancreatic Cyst | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Experimental): 1 intravenous dose followed by 1 oral dose each 12 hours (complete 3 days)
  Interventions: Drug: Placebo
- Antibiotic (Active Comparator): Ciprofloxacin 400 mg intravenous one dose followed by ciprofloxacin 500 mg oral each 12 hours (complete 3 days)
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Placebo — Evaluate usefullness of antibiotic prophylaxis
  Arms: Placebo
Drug: Ciprofloxacin — Ciprofloxacine 400 mg intravenous one dose followed by ciprofloxacine oral each 12 hours (complete 3 days)
  Arms: Antibiotic

SUMMARY:
The purpose of this study is to determine whether the use of antibiotic prophylaxis is appropriate when performing a pancreatic cyst fine needle aspiration guided by endoscopic ultrasonography.

DETAILED DESCRIPTION:
The incidence of infection after a pancreatic cyst fine needle aspiration guided by endoscopic ultrasonography (EUS-FNA) is not well known. Antibiotic prophylaxis is recommended in clinical guidelines despite the lack of evidence of its usefulness.

Our hypothesis is that the risk of infection will not be higher with placebo, and risks associated to the use of antibiotics might even increase with the use of prophylaxis.

The main objective of the project is to assess the risk of infection after the procedure and to determine whether the use of antibiotic prophylaxis is appropriate. The study is a phase IV, multicenter, double-blinded, randomized, placebo-controlled, and non-inferiority trial . We have designed a study with two parallel treatment groups. Patients will be randomized to the prophylaxis or to the placebo group. All patients will be followed for 21 days or until resolution of complications. To evaluate this primary objective with a non inferiority study, we have estimated that a total of 218 patients will be needed (109 per group) .

The main secondary objective is to assess the incidence of complications related to the use of antibiotic prophylaxis (i.e. allergic reactions, secondary infections or drug-resistant infections).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pancreatic cyst requiring EUS-FNA to complete evaluation.
* Participant is willing and able to give informed consent for participation in the study.
* Age 18 years or older.
* Ability to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

* Patients with other co-morbidities requiring antibiotic prophylaxis for endoscopic invasive procedures (such as those with cardiac valve prosthesis).
* Cystic lesion of the intestinal wall (foregut or duplication cyst).
* Use of antibiotic treatment for any other indication during the 5 days prior to the procedure.
* Pregnant woman.
* Known allergy/sensitivity to ciprofloxacin.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2014-10; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Risk of infection of a pancreatic cyst or infection related to the procedure | 21 days
  The infection can be defined as "confirmed" if there is a positive culture of the lesion content or if there is suspicion by clinical and image techniques (CT, MRI), and a positive blood culture is obtained. It will be defined as "suspected" when clinical and/or image is suggestive of cyst infection, but microbial confirmation is not obtained.

SECONDARY OUTCOMES:
Risk of fever | 21 days
  This will be measured prior to discharge. In case of clinical suspicion of bacteraemia at any moment during the follow up, blood cultures will be obtained.
secondary effects, allergic reactions, and drug resistant or secondary infections | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Guarner-Argente, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colan-Hernandez J, Sendino O, Loras C, Pardo A, Gornals JB, Concepcion M, Sanchez-Montes C, Murzi M, Andujar X, Velasquez-Rodriguez J, Rodriguez de Miguel C, Fernandez-Esparrach G, Gines A, Guarner-Argente C. Antibiotic Prophylaxis Is Not Required for Endoscopic Ultrasonography-Guided Fine-Needle Aspiration of Pancreatic Cystic Lesions, Based on a Randomized Trial. Gastroenterology. 2020 May;158(6):1642-1649.e1. doi: 10.1053/j.gastro.2020.01.025. Epub 2020 Jan 20. PMID 31972236